CLINICAL TRIAL: NCT06760559
Title: Pain Scores Following Intrarticular Injections
Brief Title: Does Pre-injection Local Anesthesia Affect Experienced Pain During Intra-articular Hip Injections.
Status: Completed | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TLV-0674-21
Record Dates: First submitted 2024-12-31; First posted 2025-01-07 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Pain; Injection; Prevention; Assessment
Keywords: pain; injection; intra-articular; expectation; compliance
MeSH Terms: conditions — Pain; Patient Compliance | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pre-injection superficial local anesthesia prior to Intra-articular corticosteroid injection
  Interventions: Procedure: Intra-articular corticosteroid injection
- Patients without pre-injection local anesthesia prior to Intra-articular corticosteroid injection
  Interventions: Procedure: Intra-articular corticosteroid injection

INTERVENTIONS:
Procedure: Intra-articular corticosteroid injection — Intra-articular hip injections with and without local anastesia and questionnaire about pain and anxiety related to the procedure was administered before and after the injection to the study and control groups.
  Other Names: Local anasthesia

SUMMARY:
Intra-articular hip injections are commonly used for diagnostic and therapeutic purposes but are often associated with patient anxiety and fear. The disparity between anticipated and experienced pain during these injections, as well as the role of pre-injection local anesthesia in pain modulation, remains unclear.

This study investigates the difference between anticipated and experienced pain during intra-articular hip injections. In addition, the study examines the impact of pre-injection local anesthesia in 60 prospectively recruited patients, some of whom received pre-injection local anesthesia while others did not. These study findings provide valuable insights into experienced pain during intra-articular hip injections, which can be applied to improve patient experiences and treatment compliance.

DETAILED DESCRIPTION:
1. Identification of patients in the outpatient clinic and completion of the questionnaires will be carried out by the principal investigator and sub-investigators in the clinic.
2. Data processing will be conducted by physicians holding an MD certification.
3. The type of study is prospective.
4. Data collection will be performed using the medical records of Tel Aviv Medical Center Hospital only, covering the years 2021 and 2022.
5. Demographic data will be collected, including gender, year of birth, age, diagnosis, indication for injection, and previous treatments. Clinical data will include underlying diseases, side of injection, complications, indications, and follow-up time.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a first-time intra-articular hip injection as indicated by an orthopedic surgeon.
* Indications for injection include:
* Diagnostic purposes (e.g., lidocaine test, arthrography)
* Therapeutic purposes (e.g., steroid injection for osteoarthritis)
* Participants must be 18 years of age or older.
* No previous hip joint injections.
* Ability to fill in the survey questionnaire.

Exclusion Criteria:

* Patients under 18 years of age.
* Patients with a known history of hypersensitivity or allergy to the injectant material (e.g., local anesthetics, steroids).
* Patients lacking the ability to sign informed consent or complete a survey questionnaire.
* Patients with previous hip joint injections, due to the potential for recalling prior pain experienced.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing first-time intra-articular hip injection as indicated by an orthopedic surgeon either for diagnostic (e.g. lidocaine test, arthrography) and/or therapeutic (steroid injection for osteoarthritis) purposes.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2022-01-02 (Actual); Study Completion 2022-01-02 (Actual)

PRIMARY OUTCOMES:
Numeric rating scales (NRS) scores | Questionnaire was given before the injection for anticipated pain evaluation and additional influencing factors on pain perception prior to injection and right after the injection for actual experienced pain.
  Numeric rating scales (NRS) scores were measured before and after an injection in both, study and control groups to determine the anticipated pain compared to experienced pain after Intra-articular hip injection with or without local anasthesia.

SECONDARY OUTCOMES:
Beck Anxiety Inventory (BAI) and fear of injections | Questionnaire was given before the injection for anticipated pain evaluation,Beck Anxiety Inventory (BAI) and additional influencing factors on pain perception prior to injection.
  Correlation of BAI scores and other injection-related factors including fear of pain, needle visualization, needle size, and prior injection experiences to pre-injection anticipated pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ehud Rath, Professor, Study Director — Tel Aviv Medical Center
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
Due to medical confidentiality